CLINICAL TRIAL: NCT04313829
Title: Impact of Pharmacist Counseling on the Health-related Quality of Life of Patients With Type 2 Diabetes Mellitus: a Cluster Randomized Controlled Study
Brief Title: Pharmacist Counseling on the Health-related Quality of Life of Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Ministry of Research, Technology and Higher Education of the Republic of Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DM-202003.01
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All patients provided written informed consent before participating in the study. The participants were administered the EQ-5D-5L questionnaire in the first month of the study, as a pre-test procedure. The patients in the control group participated in the standard Prolanis T2DM program for 6 months and were asked to fill out the questionnaire again at the 6-month time point, as a post-test procedure. The patients in the intervention group participated in the standard Prolanis T2DM program and received a 15 min face-to-face counseling session from a pharmacist once a month for 6 months. At the 6-month time point, subjects in the intervention group were asked to fill out the EQ-5D-5L questionnaire again, as a post-test procedure. Patients in the control group also received a 15 min face-to-face counseling session from a pharmacist once a month for 6 months after the intervention study was completed.
Who Masked: Care Provider
Masking Description: Cluster randomization by institution was used in this study. The four Puskesmas were randomized by asking the person in charge of the Prolanis at these centers to choose a closed envelope containing an identifier indicating the control group or the intervention group. Two Puskesmas were used as the control group and the remaining two were used as the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group received Pharmacist counseling for 15 minutes include giving standard medicine information service and explaining the validated pharmacist counseling module which contained the T2DM causes and symptoms, the reasons for the importance of therapy, the non-pharmacological and pharmacological therapies available (drug names, strengths, indications, rules of use, side effects, interactions, and storage), the purpose of controlling blood sugar levels, medications that need to be avoided, and guidelines for missed dose.
  Interventions: Behavioral: Pharmacist Counseling Intervention
- Control group (No Intervention): The control group received standard medicine information services by Pharmacists.

INTERVENTIONS:
Behavioral: Pharmacist Counseling Intervention — We used the counseling module (in the form of a guide book) for pharmacist-based counseling that had been validated regarding constructive content by an endocrinologist and a pharmacist expert in diabetes drug counseling. The module explained the T2DM causes and symptoms, the reasons for the importance of therapy, the non-pharmacological and pharmacological therapies available (drug names, strengths, indications, rules of use, side effects, interactions, and storage), the purpose of controlling blood sugar levels, medications that need to be avoided, and guidelines for missed doses. The pharmacists should explain all the content within the module in 15 minutes to each patient of the intervention group each month for 6 months. As an ethical consideration, the control group patients were given the same explanation module through pharmacist counseling after the study finished.
  Arms: Intervention group

SUMMARY:
The quality of life (QoL) of patients with type 2 diabetes mellitus (T2DM) is a measure of the successful outcomes of therapy. The program of management of chronic diseases "Program Pengelolaan Penyakit Kronis" (Prolanis) among patients with hypertension and T2DM is a new strategy of the Badan Penyelenggara Jaminan Sosial (BPJS), which is the Indonesian national health insurance system. The impact of pharmacist counseling interventions on health-related QoL (HRQoL) was analyzed in Prolanis T2DM patients.

DETAILED DESCRIPTION:
A cluster randomized controlled trial that was designed to include two groups (control (n = 111) and intervention (n = 109) groups), and pre- and post-test procedures were conducted. The participants were Prolanis T2DM patients who attended four primary health-care centers (Puskesmas) in Makassar City, South Sulawesi, Indonesia from August 2017 to August 2018. The intervention group received systematic counseling for 6 months. The data were collected using the Bahasa Indonesia version of the European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire and were analyzed using EQ-5D preference weight for each health state with the Indonesian EQ-5D-5L value Set. Furthermore, the EQ-5D index and the EQ-5D VAS score were calculated and HbA1c levels were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Registration in the Prolanis at BPJS Makassar City,
* Age between 20 and 65 years,
* HbA1c level ≥6.5%, and
* Willingness to participate in research by signing an informed consent (for all T2DM patients with or without comorbidities)

Exclusion Criteria:

* Irregular control schedules,
* Incomplete medical record data,
* Circumstances that did not allow filling out the questionnaires (e.g., inability to speak, see, or hear)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of Quality of Life (QoL) using the Euro Quality of Life 5 Dimension 5 Level (EQ-5D-5L) questionnaire | 6 months
  The QoL of Prolanis T2DM patients was measured using the Euro Quality of Life 5 Dimension 5 Level (EQ-5D-5L) questionnaire.
  The EQ-5D-5L questionnaire consists of two parts: a descriptive system and a Visual Analogue Scale (VAS).
  The descriptive system describes the health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients who reported problems were then categorized into two categories, a "has no problem" category (health state code of 1) and "has problem" category (health state code of 2-5) for each level of each dimension.
  The second part of the EQ-5D-5L questionnaire is the EQ-VAS, which is a thermometer-like scale (ranging from 0 to 100) that reflects the patient's health in general. EQ-VAS represents the patient perspective, where zero indicates the worst imaginable health state and 100 reflects the best imaginable health state.

SECONDARY OUTCOMES:
Measurement of HbA1c | 6 months
  Measurement of HbA1c was done over a period of 2-4 months. In addition, HbA1c was also be considered compatible with therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Fajriansyah Fajriansyah, Master, Principal Investigator — Faculty of Pharmacy Universitas Padjadjaran Bandung
Locations (4):
- Indonesia (4):
  - Puskesmas Antang, Makassar, South Sulawesi
  - Puskesmas Batua, Makassar, South Sulawesi
  - Puskesmas Jongaya, Makassar, South Sulawesi
  - Puskesmas Tamalanrea, Makassar, South Sulawesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Purba FD, Hunfeld JAM, Iskandarsyah A, Fitriana TS, Sadarjoen SS, Ramos-Goni JM, Passchier J, Busschbach JJV. The Indonesian EQ-5D-5L Value Set. Pharmacoeconomics. 2017 Nov;35(11):1153-1165. doi: 10.1007/s40273-017-0538-9. PMID 28695543
- [Background] Agborsangaya CB, Lau D, Lahtinen M, Cooke T, Johnson JA. Health-related quality of life and healthcare utilization in multimorbidity: results of a cross-sectional survey. Qual Life Res. 2013 May;22(4):791-9. doi: 10.1007/s11136-012-0214-7. Epub 2012 Jun 9. PMID 22684529
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Result] Steinsbekk A, Rygg LO, Lisulo M, Rise MB, Fretheim A. Group based diabetes self-management education compared to routine treatment for people with type 2 diabetes mellitus. A systematic review with meta-analysis. BMC Health Serv Res. 2012 Jul 23;12:213. doi: 10.1186/1472-6963-12-213. PMID 22824531
- [Result] Megari K. Quality of Life in Chronic Disease Patients. Health Psychol Res. 2013 Sep 23;1(3):e27. doi: 10.4081/hpr.2013.e27. eCollection 2013 Sep 24. PMID 26973912
- [Result] Kjeldsen LJ, Bjerrum L, Dam P, Larsen BO, Rossing C, Sondergaard B, Herborg H. Safe and effective use of medicines for patients with type 2 diabetes - A randomized controlled trial of two interventions delivered by local pharmacies. Res Social Adm Pharm. 2015 Jan-Feb;11(1):47-62. doi: 10.1016/j.sapharm.2014.03.003. Epub 2014 Apr 12. PMID 24798710
- [Result] Nichols GA, Rosales AG, Kimes TM, Tunceli K, Kurtyka K, Mavros P. The Change in HbA1c Associated with Initial Adherence and Subsequent Change in Adherence among Diabetes Patients Newly Initiating Metformin Therapy. J Diabetes Res. 2016;2016:9687815. doi: 10.1155/2016/9687815. Epub 2016 Aug 7. PMID 27579326
- [Result] van Eikenhorst L, Taxis K, van Dijk L, de Gier H. Pharmacist-Led Self-management Interventions to Improve Diabetes Outcomes. A Systematic Literature Review and Meta-Analysis. Front Pharmacol. 2017 Dec 14;8:891. doi: 10.3389/fphar.2017.00891. eCollection 2017. PMID 29311916
- [Result] Gusmai Lde F, Novato Tde S, Nogueira Lde S. [The influence of quality of life in treatment adherence of diabetic patients: a systematic review]. Rev Esc Enferm USP. 2015 Oct;49(5):839-46. doi: 10.1590/S0080-623420150000500019. Portuguese. PMID 26516756